CLINICAL TRIAL: NCT00295698
Title: Studies on the Interaction Between HIV Infection, Lymphatic Filariasis and Diethylcarbamazine
Brief Title: Interaction Between HIV and Lymphatic Filariasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DBL -Institute for Health Research and Development (Other)
Collaborators: Danish Council for Development Research (Other); The AIDS Foundation, Denmark (Other); The Wedell-Wedellsborg Foundation, Denmark (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RUF 91088
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2006-02-24 (Estimated); Status verified 2006-02

CONDITIONS: HIV Infection; Lymphatic Filariasis
Keywords: HIV; Lymphatic filariasis; Diethylcarbamazine; Interaction; Tanzania
MeSH Terms: conditions — HIV Infections; Elephantiasis, Filarial | interventions — Diethylcarbamazine

INTERVENTIONS:
Drug: Diethylcarbamazine

SUMMARY:
The impact of lymphatic filariasis (LF) on HIV is assessed by measuring HIV viral load before and after DEC treatment of filariasis in double-infected individuals. The impact of HIV on lymphatic filariasis is assessed by measuring the success of DEC treatment on W. bancrofti antigenaemia and microfilaraemia in double-infected individuals. The effect of DEC treatment in individuals with lymphatic filariasis and/or HIV is assessed by measuring the pre- and post-treatment level of HIV viral load, immunological responses and micronutritional parameters, including antioxidants and markers of oxidative stress, in single- or double-infected individuals. The study is carried out as an anonymous, unlinked and double-blind placebo controlled study with cross-over design. The study groups comprise: 1) 18 double-infected individuals (HIV+/LF+), 2) 16 HIV infected individuals (HIV+/LF-) and 3) 25 individuals with lymphatic filariasis (HIV-/LF+). Based on stratified, blocked randomisation the study participants receive DEC treatment or placebo. Pre- and post-treatment (1 week, 12 weeks and 24 weeks post-treatment) blood samples are collected and analysed for HIV viral load, CD4+ T cell count, distinctive Th1 and Th2 cytokines, circulating filarial antigens (CFA), micronutrient status, antioxidant enzymes and markers of oxidative stress. After 12 weeks the study participants get the opposite treatment and post-treatment blood samples are collected four times with the same intervals as above.

DETAILED DESCRIPTION:
Previous studies on the interaction between HIV and helminth infections have indicated that HIV may have a negative impact on helminth infections and vice versa, and there is evidence that treatment of chronic helminth infections in HIV infected individuals can delay the progression of HIV. These interactions may be related to changes in the immunological responsiveness or through an effect on reactive oxygen compounds resulting in oxidative stress. Oxidative stress may be a neglected determinant for progression of lymphatic filariasis and may also impair immune functions and lead to increased HIV replication through activation of nuclear transcription factors. The present study examines the three-way interaction between HIV infection, lymphatic filariasis caused by the helminth parasite W. bancrofti and the drug diethylcarbamazine (DEC). DEC is an important drug for treatment of lymphatic filariasis and previous findings indicate that DEC may also have an effect on retroviral infections.

The impact of lymphatic filariasis (LF) on HIV is assessed by measuring HIV viral load before and after DEC treatment of filariasis in double-infected individuals. The impact of HIV on lymphatic filariasis is assessed by measuring the success of DEC treatment on W. bancrofti antigenaemia and microfilaraemia in double-infected individuals. The effect of DEC treatment in individuals with lymphatic filariasis and/or HIV is assessed by measuring the pre- and post-treatment level of HIV viral load, immunological responses and micronutritional parameters, including antioxidants and markers of oxidative stress, in single- or double-infected individuals. The study is carried out as an anonymous, unlinked and double-blind placebo controlled study with cross-over design. The study groups comprise: 1) 18 double-infected individuals (HIV+/LF+), 2) 16 HIV infected individuals (HIV+/LF-) and 3) 25 individuals with lymphatic filariasis (HIV-/LF+). Based on stratified, blocked randomisation the study participants receive DEC treatment or placebo. Pre- and post-treatment (1 week, 12 weeks and 24 weeks post-treatment) blood samples are collected and analysed for HIV viral load, CD4+ T cell count, distinctive Th1 and Th2 cytokines, circulating filarial antigens (CFA), micronutrient status, antioxidant enzymes and markers of oxidative stress. After 12 weeks the study participants get the opposite treatment and post-treatment blood samples aree collected four times with the same intervals as above.

If treatment of coexisting helminth infections, including lymphatic filariasis, delays the progression of HIV, such treatment may be an important measure to alleviate the effect of the AIDS epidemic in Africa and other areas where HIV and helminths coexist. For lymphatic filariasis in particular such information will be of high significance in the strategic planning by decision-makers within the ongoing international efforts for control of lymphatic filariasis.

ELIGIBILITY:
Inclusion Criteria:

One of the three following conditions:

1. Positivity for antibodies to HIV-1 or HIV-2
2. Positivity for circulating filarial antigen from W. bancrofti
3. Positivity for both HIV antibodies and W.bancrofti circulating antigens

Exclusion Criteria:

1. AIDS
2. Hydrocele
3. Lymphoedema
4. Elephantiasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-08; Study Completion 2002-11

CONTACTS AND LOCATIONS:
Overall Officials: Nina O Nielsen, Ms.c, Principal Investigator — DBL -Institute for Health Research and Development